CLINICAL TRIAL: NCT06689748
Title: Training Curriculum For Physicians Involved With Airway Management In Critically Ill Patients: A Delphi Study
Brief Title: Curriculum for Airway Skills in Critically Ill Adults: a Delphi Evaluation
Acronym: CASCADE
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kunal Karamchandani, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-1102
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Airway Management; Tracheal Intubation; Critical Illness; Training
Keywords: Airway management; Tracheal intubation; Training curriculum; Critical illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experts: Airway management experts The Steering Committee selected Experts from across the globe based on pre-defined criteria and will conduct iterative Delphi rounds to generate consensus among the experts.
  Interventions: Other: Delphi procedure

INTERVENTIONS:
Other: Delphi procedure — The study involves generating consensus statements by experts on the training requirements for physicians involved with airway management in critically ill patients using a Delphi process.

SUMMARY:
This study using a Delphi methodology, and involving international experts, will help define a training curriculum for physicians involved with airway management in critically ill patients.

DETAILED DESCRIPTION:
Airway management in critically ill patients is associated with significant morbidity and mortality. In an international Delphi study, the need for a training curriculum for airway management in critically Ill patients was identified. While attempts have been made to collaborate and define the training requirements in this field, further clarity is needed. In order to define the essential components of the training curriculum for airway management in critically ill patients, we plan to conduct an Delphi study involving a diverse group of international experts from various specialities, involved with airway management in critically ill patients.

The Delphi process is a well-established methodology to generate consensus on a particular topic using the "collective intelligence" of panel members.5,6 The steering committee members performed a literature search on the available evidence, including existing curriculum for airway management, drafted the initial statements, and will conduct iterative Delphi rounds to generate consensus among the experts. The Steering Committee members will not participate in the Delphi surveys themselves. The study findings will be reported according to the ACCORD criteria.

Steps of the Delphi process Step 1: Establishing a preliminary list of broad domains A focused literature review will be performed by the members of the SC and based on their input, the steering committee will identify broad domains, which will be used to draft statements for Round one of the Delphi process.

Step 2: Preparation of the Delphi Round One Survey The list of questions related to the above-mentioned domains will be sent to the Experts as a Delphi questionnaire. The anonymity of the Experts will be maintained until the end of the Delphi rounds. The Experts would be requested to answer questions related to training curriculum based on their experience and knowledge of the subject. The questions will be multiple choice or in the form of a 7-point Likert scale (strongly agree, agree, somewhat agree, neither agree nor disagree, somewhat disagree, disagree, strongly disagree). The experts can also provide their opinion on addition, deletion on questions or choices through free-text. The responses of experts will be collated during the analysis of results and shared in the following survey as controlled feedback.

Step 3: Subsequent Delphi Rounds The steering committee will review the results of round one. The statements listed will be modified, deleted, or added if found ambiguous based on the feedback and comments of the results. The remaining statements will be continued in the subsequent rounds until the stability of the responses is achieved. The cumulative results of round two will be presented to experts along with anonymized comments, and the survey process will be repeated with the modified questionnaire. The Delphi rounds will be continued until the desired consensus and stability is achieved for statements. .

Step 4: Final Consensus Only the statements that achieved consensus and stability will be used develop consensus statements. The results of the last stable round will be used to issue the consensus statements related to the above-mentioned domains. The results of the final survey, consensus statements, and the manuscript will be circulated among the experts for approval before submission for publication.

Statistical analysis

A descriptive analysis of the preliminary survey will be performed. For the Delphi process, stability will be checked by non-parametric chi-square (χ2) tests or Kruskal-Wallis test from round two onwards. A statement is said to be stable if p-value is > 0.05 for two consecutive rounds Consensus will be considered reached when a statement achieves >=75% of votes for multiple-choice questions and likert-scale statements. A statement will be continued in the questionnaire round until response stability is achieved. Consensus statements will be considered as those that generate both consensus and stability.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical expertise in airway management of critically ill patients
2. Educators with expertise in teaching and training in airway management of critically ill patients.
3. At least one publication and/or research project related to airway management in critically ill patients.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A diverse (specialty, geography, sex, country income) group of physicians meeting all of the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Consensus statements | Through study completion, an average of 12 months
  Consensus amongst the expert panel regarding training requirements for physicians involved with airway management in critically ill patients will be achieved using Delphi method which includes iterative rounds of questions.
  Consensus will be considered reached when a statement achieves >=75% of votes for multiple-choice questions and likert-scale statements.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT06689748/Prot_SAP_000.pdf